CLINICAL TRIAL: NCT03879720
Title: Comparison of Standard Endotracheal Intubation [SEI] and Endoscope Assisted Endotracheal Intubation [EAE]
Brief Title: Comparison of Standard and Endoscope Assisted Endotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Subhas Banerjee, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47089
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Biliary Tract Diseases; Pancreatic Diseases
Keywords: ERCP; Endoscopic Procedures; Anesthesia
MeSH Terms: conditions — Biliary Tract Diseases; Pancreatic Diseases

STUDY DESIGN:
Intervention Model Description: Randomization to standard endotracheal intubation or endoscopist-facilitated endotracheal intubation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Endotracheal Intubation (SEI) (Active Comparator): the patient will be positioned supine on the gurney for intubation, with eventual position in the standard semi-prone ERCP position on the fluoroscopy table. Anesthesiologist-determined doses of Fentanyl, Versed, Propofol and Succinylcholine will be administered per standard of care and intubation will be accomplished by direct laryngoscopy or glidescope, with confirmation of endotracheal tube placement by auscultation.
  Interventions: Procedure: Endoscope assisted endotracheal intubation [EAEI]
- Endoscope assisted endotracheal intubation [EAEI] (Experimental): the patients will position themselves in the semi-prone position on the fluoroscopy table. Anesthesiologist-determined doses of Fentanyl, Versed and Propofol will be administered per standard of care. Succinylcholine will not be administered and therefore the patient will not be paralyzed. The endotracheal tube will be positioned on the mid-distal aspect of the ultra-slim endoscope and the ultra-slim endoscope will then be advanced into the trachea under direct endoscopic visualization to the level of the carina. The anesthesiologist will then advance the endotracheal tube over the endoscope into the trachea, and its position above the carina will be simultaneously confirmed endoscopically with the ultra-slim endoscope.
  Interventions: Procedure: Endoscope assisted endotracheal intubation [EAEI]

INTERVENTIONS:
Procedure: Endoscope assisted endotracheal intubation [EAEI] — Endoscope assisted endotracheal intubation [EAEI] performed by anesthesiologist with endoscopist assistance.
  Other Names: Standard Endotracheal Intubation [SEI]

SUMMARY:
Comparison of standard endotracheal intubation and endoscopist-facilitated endotracheal intubation

DETAILED DESCRIPTION:
Endoscopic Retrograde Cholangiopancreatography (ERCP) procedures are typically performed using general anesthesia. During anesthesia, the anesthesiologist inserts a breathing tube (endotracheal tube) into the patient's wind pipe (trachea) and a machine helps the patient breathe (mechanical ventilation) while they are unconscious. The breathing tube is inserted with a patient laying on his/her back using a rigid metallic device (laryngoscope) to guide tube placement. The unconscious patient is then moved from the portable bed onto the X-ray table by nursing staff. The patient also has to be turned to lie on their stomach on the X-ray table for the procedure. This standard approach carries a small risk of patient injury during breathing tube placement as well as while moving and turning the unconscious patient onto the X-ray table.

At our endoscopy unit, endoscopists have, on several occasions, used a slim gastroscope to place the breathing tube under direct visualization in patients who are already positioned on their stomach for ERCP. This approach is rapid and has been uniformly successful and safe.

We hypothesize that this endoscopist-facilitated intubation approach may expedite the procedure and minimize ergonomic strain for staff during patient repositioning while minimizing patient injury during breathing tube placement and repositioning. This study seeks to formally compares the two approaches for placement of a breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ERCP at Stanford University Medical Center

Exclusion Criteria:

* Unable to consent
* Contra-indication to general anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to Procedure Start | up to 1 hour
  Time from patient entry into procedure room to insertion of endoscope/start of procedure

SECONDARY OUTCOMES:
Intubation Time (time from 'ready to intubate', to 'tube confirmation') | up to 1 hour
  Endoscopy documentation
Patient positioning time | up to 1 hour
  Recorded in endoscopy suite
Staff required for patient positioning | up to 20 minutes
  Recorded in endoscopy suite, # of staff
Staff survey/assessment of ergonomic strain | up to 1 hour
  Staff reporting of ergonomic strain encountered during the procedure scale of 1-5 to rate ergonomic strain,
Need for special positioning equipment | up to 20 minutes
  Documented based on procedure room observation, list of equipment
Hypoxia (nadir O2 sat and duration), Arrhythmia, Hypotension | up to 20 minutes
  Evaluation of hypoxia during intubation
Time from removal of GI endoscope to exit from procedure room | up to 60 minutes
  Documented in endoscopy suite
Tooth/oropharyngeal trauma, skin/musculoskeletal trauma | up to 24 hours post-procedure
  Evaluation of oropharyngeal trauma and skin/musculoskeletal complaints following intubation, rating scale (0-5 to rate damage)
Materials and facility fees | up to 24 hours post-procedure
  assessment of cost associated with procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barakat MT, Angelotti T, Ghosh S, Banerjee S. Prospective randomized comparison of endoscopist-facilitated endotracheal intubation and standard intubation for ERCP. Gastrointest Endosc. 2023 Sep;98(3):441-447. doi: 10.1016/j.gie.2023.02.032. Epub 2023 Mar 5. PMID 36878302